CLINICAL TRIAL: NCT00193570
Title: A Phase I Study of Topotecan in Combination With Docetaxel in Patients With Refractory and/or Advanced Solid Tumors
Brief Title: Topotecan in Combination With Docetaxel in Refractory and/or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry); Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 34; 104864652
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Topotecan; Docetaxel

INTERVENTIONS:
Drug: Topotecan
Drug: Docetaxel

SUMMARY:
This phase I study will characterize the safety, tolerability, and maximum tolerated dose and dose-limiting toxicity of weekly bolus Topotecan when administered in combination with to different dosing regimens of docetaxel. We will also evaluate any anti-tumor activity of the combination regimen.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

For ever 2 patients treated, 1 will receive treatment A (Paclitaxel + Carboplatin + Gemcitabine) and 1 will receive treatment B (Gemcitabine + Vinorelbine). The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

Upon determination of eligibility, patients will be receive:

* Docetaxel + Topotecan

In order to determine the most appropriate dosing regimen to progress into future phase II trials, two different dosing schedules of Topotecan and docetaxel will be utilized.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Adult > 18 years of age
* ECOG performance status 0 or 1
* Received 3 or less chemotherapy regimens in the metastatic setting
* Adequate bone marrow, liver and kidney function
* Prior brain metastases must be inactive and asymptomatic
* No previous treatment with Topotecan or docetaxel
* Understand the nature of the study and give written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Moderate or severe peripheral neuropathy
* Active concurrent infection or serious underlying medical condition
* Known HIV positivity
* Pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-02; Primary Completion 2004-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose of drug combination

SECONDARY OUTCOMES:
Response rates

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, MD, Principal Investigator — SCRI Development Innovations, LLC